CLINICAL TRIAL: NCT06593951
Title: Registry and Natural History Study for Progressive Myoclonus Epilepsy Type 1 (EPM1)
Acronym: EPM1
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Epilepsy Foundation (Other)
Responsible Party: Principal Investigator, Darius Ebrahimi-Fakhari, Darius Ebrahimi-Fakhari, MD, PhD, Boston Children's Hospital
Other Study IDs: IRB-P00048807
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Progressive Myoclonus Epilepsy Type 1; EPM1; CSTB-related Disease; Myoclonus Epilepsies, Progressive; Unverricht-Lundborg Disease; Progressive Epilepsy and/or Ataxia With Myoclonus as a Major Feature; PME; Progressive Myoclonus-Epilepsies
Keywords: Myoclonus; Progressive Myoclonus; CSTB; Non-epileptic action-induced myoclonus; Non-epileptic stimulus-induced myoclonus; Cerebellar disfunction; EPM1
MeSH Terms: conditions — Myoclonic Epilepsies, Progressive; Unverricht-Lundborg Syndrome; Myoclonus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood and / or urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Registry and Natural History Study for Progressive Myoclonus Epilepsy Type 1 (EPM1) is focused on gathering longitudinal clinical data as well as biological samples (blood and/or urine) from male and female patients, of all ages, who have a molecular diagnosis of EPM1or CSTB-null-related disease. Currently, there are no therapies that halt disease progression in any CSTB-related diseases, highlighting the urgency for translational research into this condition. The primary objective of the registry is to determine the natural history and genotype-phenotype correlations of disease-causing variants in EPM1 and CSTB-null-related disease.

DETAILED DESCRIPTION:
Progressive myoclonus-epilepsies (PME) are severe epilepsies that insinuate into the lives of previously healthy children or young adults, irrevocably intensify, and become intractable. Progressive Myoclonic Epilepsy type 1 (EPM1), also known as Unverricht-Lundborg disease (ULD), is the prototypical and most common PME. It is caused by bi-allelic variants in the CSTB gene. The phenotypic spectrum of EPM1 is broad and reflects the amount of residual CSTB protein function in an individual. Individuals with classic EPM1 typically develop seizures between 6-16 years of age, followed by progressive non-epileptic action- and stimulus-induced myoclonus, ataxia, and cerebellar dysfunction with speech and swallowing impairment. These individuals generally have one or both CSTB variants partially functional. On the severe end of the spectrum are patients with a complete loss of the CSTB protein due to bi-allelic null variants.

The characterization of disease progression and biomarker discovery are necessary to define clinically meaningful endpoints for future interventional trials and to meet regulatory requirements for phase 1/2 and later-stage trials.

As an ultra-rare disease, patients with EPM1 are dispersed across the United States, making on-site visits for natural history studies burdensome to families. In this study, we will overcome this obstacle by adapting a remote- assessment-driven natural history study with clinical, electrophysiological, and biochemical biomarkers. The proposed study will delineate the natural history and evolution of myoclonus as a key disease feature in EPM1 and CSTB-related disease, will create a biobank for biospecimen, and will assess health-related quality of life. This approach will further clinical trial readiness for EPM1-related disease.

Specifically, the objectives of this protocol are to:

1. Determine the natural history and genotype-phenotype correlations of disease-causing variants in EPM1-related disease.
2. Facilitate an early diagnosis, enable counseling with anticipatory guidance of affected families and help define clinically meaningful endpoints for future interventional traits.

Specific aims include:

1. Perform longitudinal Unified Myoclonus Rating Scale (UMRS) assessments and clinical interviews via video-teleconference with study participants to track functional impairment and disease progression.
2. Establish a biobank for samples from participants with CSTB mutations, including EPM1 and CSTB-null disease, enabling quantitative profiling of biochemical biomarkers.
3. Conduct a health-related quality of life survey about participants with EPM1 and CSTB-null disease to understand the impact on patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Molecular diagnosis of EPM1-related disease
* Access to web-based communication, including video-teleconference
* Permanent address in the United States

Exclusion Criteria:

* Not having such a diagnosis of EPM1-related disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of male and female patients of all ages with a clinical and molecular diagnosis of EPM1-related disease.
  The initial phase of this study will enroll a minimum of 10 individuals with EPM1-related disease. A total of 200 individuals may be entered in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Unified Myoclonus Rating Scale (UMRS) | 5 years
  Perform longitudinal Unified Myoclonus Rating Scale (UMRS) assessments and clinical interviews via video-teleconference in EPM1 patients to track functional impairment and disease progression.
Creation of Biorepository | 5 years
  Establish a biobank for patients with CSTB mutations, including EPM1 and CSTB-null disease, enabling quantitative profiling of biochemical biomarkers.
Assess Health-Related Quality of Life | 5 years
  Conduct a health-related quality of life survey on EPM1 and CSTB-null disease patients to understand the priorities of and impact on patients and caregivers.

SECONDARY OUTCOMES:
Establish clinical trial readiness | 5 years
  To facilitate an early diagnosis, enable counseling and anticipatory guidance of affected families and help define clinically meaningful endpoints for future interventional trials.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Childrens Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rissanen SM, Hypponen J, Silvennoinen K, Saisanen L, Karjalainen PA, Mervaala E, Kalviainen R. Wearable monitoring of positive and negative myoclonus in progressive myoclonic epilepsy type 1. Clin Neurophysiol. 2021 Oct;132(10):2464-2472. doi: 10.1016/j.clinph.2021.06.026. Epub 2021 Jul 30. PMID 34454274
- [Background] Joensuu T, Lehesjoki AE, Kopra O. Molecular background of EPM1-Unverricht-Lundborg disease. Epilepsia. 2008 Apr;49(4):557-63. doi: 10.1111/j.1528-1167.2007.01422.x. Epub 2007 Nov 19. PMID 18028412
- [Background] Hadady L, Klivenyi P, Fabo D, Beniczky S. Real-world user experience with seizure detection wearable devices in the home environment. Epilepsia. 2023 Dec;64 Suppl 4:S72-S77. doi: 10.1111/epi.17189. Epub 2022 Feb 23. PMID 35195898
- [Background] Hainque E, Vidailhet M, Cozic N, Charbonnier-Beaupel F, Thobois S, Tranchant C, Brochard V, Glibert G, Drapier S, Mutez E, Doe De Maindreville A, Lebouvier T, Hubsch C, Degos B, Bonnet C, Grabli D, Legrand AP, Meneret A, Azulay JP, Bissery A, Zahr N, Clot F, Mallet A, Dupont S, Apartis E, Corvol JC, Roze E. A randomized, controlled, double-blind, crossover trial of zonisamide in myoclonus-dystonia. Neurology. 2016 May 3;86(18):1729-35. doi: 10.1212/WNL.0000000000002631. Epub 2016 Apr 6. PMID 27053715
- [Background] Mullard A. NfL makes regulatory debut as neurodegenerative disease biomarker. Nat Rev Drug Discov. 2023 Jun;22(6):431-434. doi: 10.1038/d41573-023-00083-z. No abstract available. PMID 37198334
- [Background] Nasseri M, Pal Attia T, Joseph B, Gregg NM, Nurse ES, Viana PF, Worrell G, Dumpelmann M, Richardson MP, Freestone DR, Brinkmann BH. Ambulatory seizure forecasting with a wrist-worn device using long-short term memory deep learning. Sci Rep. 2021 Nov 9;11(1):21935. doi: 10.1038/s41598-021-01449-2. PMID 34754043
- [Background] Okuneva O, Korber I, Li Z, Tian L, Joensuu T, Kopra O, Lehesjoki AE. Abnormal microglial activation in the Cstb(-/-) mouse, a model for progressive myoclonus epilepsy, EPM1. Glia. 2015 Mar;63(3):400-11. doi: 10.1002/glia.22760. Epub 2014 Oct 18. PMID 25327891
- [Background] O'Brien A, Marshall CR, Blaser S, Ray PN, Yoon G. Severe neurodegeneration, progressive cerebral volume loss and diffuse hypomyelination associated with a homozygous frameshift mutation in CSTB. Eur J Hum Genet. 2017 Jun;25(6):775-778. doi: 10.1038/ejhg.2017.39. Epub 2017 Apr 5. PMID 28378817
- [Background] Mancini GM, Schot R, de Wit MC, de Coo RF, Oostenbrink R, Bindels-de Heus K, Berger LP, Lequin MH, de Vries FA, Wilke M, van Slegtenhorst MA. CSTB null mutation associated with microcephaly, early developmental delay, and severe dyskinesia. Neurology. 2016 Mar 1;86(9):877-8. doi: 10.1212/WNL.0000000000002422. Epub 2016 Feb 3. No abstract available. PMID 26843564
- [Background] Lehesjoki AE, Koskiniemi M, Sistonen P, Miao J, Hastbacka J, Norio R, de la Chapelle A. Localization of a gene for progressive myoclonus epilepsy to chromosome 21q22. Proc Natl Acad Sci U S A. 1991 May 1;88(9):3696-9. doi: 10.1073/pnas.88.9.3696. PMID 1673790
- [Background] Kalviainen R, Genton P, Andermann E, Andermann F, Magaudda A, Frucht SJ, Schlit AF, Gerard D, de la Loge C, von Rosenstiel P. Brivaracetam in Unverricht-Lundborg disease (EPM1): Results from two randomized, double-blind, placebo-controlled studies. Epilepsia. 2016 Feb;57(2):210-21. doi: 10.1111/epi.13275. Epub 2015 Dec 15. PMID 26666500
- [Background] Houseweart MK, Pennacchio LA, Vilaythong A, Peters C, Noebels JL, Myers RM. Cathepsin B but not cathepsins L or S contributes to the pathogenesis of Unverricht-Lundborg progressive myoclonus epilepsy (EPM1). J Neurobiol. 2003 Sep 15;56(4):315-27. doi: 10.1002/neu.10253. PMID 12918016
- [Background] Gumusgoz E, Kasiri S, Verma M, Wu J, Villarreal Acha D, Marriam U, Fyffe-Maricich S, Lin A, Chen X, Gray SJ, Minassian BA. CSTB gene replacement improves neuroinflammation, neurodegeneration and ataxia in murine type 1 progressive myoclonus epilepsy. Gene Ther. 2024 May;31(5-6):234-241. doi: 10.1038/s41434-023-00433-x. Epub 2023 Dec 22. PMID 38135787
- [Background] Frucht SJ, Louis ED, Chuang C, Fahn S. A pilot tolerability and efficacy study of levetiracetam in patients with chronic myoclonus. Neurology. 2001 Sep 25;57(6):1112-4. doi: 10.1212/wnl.57.6.1112. PMID 11571347
- [Background] Frucht SJ, Leurgans SE, Hallett M, Fahn S. The Unified Myoclonus Rating Scale. Adv Neurol. 2002;89:361-76. No abstract available. PMID 11968461
- [Background] Di Matteo F, Pipicelli F, Kyrousi C, Tovecci I, Penna E, Crispino M, Chambery A, Russo R, Ayo-Martin AC, Giordano M, Hoffmann A, Ciusani E, Canafoglia L, Gotz M, Di Giaimo R, Cappello S. Cystatin B is essential for proliferation and interneuron migration in individuals with EPM1 epilepsy. EMBO Mol Med. 2020 Jun 8;12(6):e11419. doi: 10.15252/emmm.201911419. Epub 2020 May 7. PMID 32378798
- [Background] Daura E, Tegelberg S, Yoshihara M, Jackson C, Simonetti F, Aksentjeff K, Ezer S, Hakala P, Katayama S, Kere J, Lehesjoki AE, Joensuu T. Cystatin B-deficiency triggers ectopic histone H3 tail cleavage during neurogenesis. Neurobiol Dis. 2021 Aug;156:105418. doi: 10.1016/j.nbd.2021.105418. Epub 2021 Jun 5. PMID 34102276
- [Background] Crespel A, Ferlazzo E, Franceschetti S, Genton P, Gouider R, Kalviainen R, Korja M, Lehtinen MK, Mervaala E, Simonato M, Vaarmann A. Unverricht-Lundborg disease. Epileptic Disord. 2016 Sep 1;18(S2):28-37. doi: 10.1684/epd.2016.0841. PMID 27582036
- [Background] Assenza G, Nocerino C, Tombini M, Di Gennaro G, D'Aniello A, Verrotti A, Marrelli A, Ricci L, Lanzone J, Di Lazzaro V, Bilo L, Coppola A. Perampanel Improves Cortical Myoclonus and Disability in Progressive Myoclonic Epilepsies: A Case Series and a Systematic Review of the Literature. Front Neurol. 2021 Mar 24;12:630366. doi: 10.3389/fneur.2021.630366. eCollection 2021. PMID 33841303
- [Background] Alecu JE, Saffari A, Ziegler M, Jordan C, Tam A, Kim S, Leung E, Szczaluba K, Mierzewska H, King SD, Santorelli FM, Yoon G, Trombetta B, Kivisakk P, Zhang B, Sahin M, Ebrahimi-Fakhari D. Plasma Neurofilament Light Chain Is Elevated in Adaptor Protein Complex 4-Related Hereditary Spastic Paraplegia. Mov Disord. 2023 Sep;38(9):1742-1750. doi: 10.1002/mds.29524. Epub 2023 Jul 22. PMID 37482941